CLINICAL TRIAL: NCT02403271
Title: A Multi-Center Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Combination With Durvalumab (MEDI4736), in Subjects With Relapsed or Refractory Solid Tumors
Brief Title: A Multi-Center Study of Ibrutinib in Combination With MEDI4736 in Subjects With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1135-CA
Record Dates: First submitted 2015-02-27; First posted 2015-03-31 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Non-Small Cell Lung Cancer; Breast Cancer; Pancreatic Cancer
Keywords: Pharmacyclics; PCYC; Ibrutinib; Durvalumab (MEDI4736); Relapsed Refractory Solid Tumor; Non-Small Cell Lung Cancer; NSCLC; Squamous; Squamous NSCLC; Squamous Non-Small Cell Lung Cancer; Immunotherapy; IMBRUVICA®; Tumor Immunotherapy; Anti-PD-L1; Lung Cancer; Breast Cancer; Triple Negative; HER2 Positive; HER2 + Breast Cancer; Pancreatic Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Pancreatic Neoplasms; Lung Neoplasms | interventions — ibrutinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1b (Experimental): In the Phase 1b (safety portion) of the study, a starting dose of 560 mg of ibrutinib and 10 mg/kg of MEDI4736 will be explored and will follow a 6+3 dose de-escalation design and will include a sentinel participant which will have a 3-day observation period prior to dosing of subsequent participants. Participants with one of the following three tumor types will be eligible for enrollment: NSCLC (adenocarcinoma and squamous-cell carcinoma), Breast cancer (triple-negative and HER2-positive cancer), and Pancreatic cancer (adenocarcinoma).
  Interventions: Drug: Ibrutinib; Drug: Durvalumab
- Phase 2 (Experimental): Participants with one of three solid tumor types (Stage III/IV) will be enrolled in the Phase 2 portion of this protocol: NSCLC (adenocarcinoma and squamous-cell carcinoma), Breast cancer (triple-negative and HER2-positive cancer), and Pancreatic cancer (adenocarcinoma) and treated at the R2PD of ibrutinib and durvalumab determined in Phase 1b. An interim analysis will be performed to evaluate the response and the safety profile, and the study may be discontinued based on the interim efficacy and/or safety results.
  Interventions: Drug: Ibrutinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Ibrutinib — BTK Inhibitor
  Other Names: PCI-32765
Drug: Durvalumab — Anti PDL-1
  Other Names: MEDI4736

SUMMARY:
This is a Phase 1b/2, multi-center study to assess the safety and efficacy of ibrutinib in combination with durvalumab (MEDI4736) in participants with relapsed or refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed: Non-small cell lung cancer (NSCLC, adenocarcinoma or squamous-cell carcinoma), Breast Cancer (HER2 positive or triple negative), Pancreatic Cancer (adenocarcinoma)
2. Relapsed or refractory disease (Stage III or IV): NSCLC or pancreatic cancer must have failed at least 1 prior treatment. Breast cancer must have failed at least 2 prior treatments.
3. Measurable lesion by RECIST 1.1
4. Adequate hematologic function:

   * ANC >1500 cells/mm3
   * Platelet count >100,000 cells/mm3
   * HGB >9.0 g/dL
5. Adequate hepatic and renal function:

   * AST and ALT ≤2.5 x ULN for subjects without liver metastases and ≤3.5 x ULN for subjects with liver metastases
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
   * Creatinine ≤2.0 x ULN and Creatinine Clearance ≥40 mL/min (Cockcroft-Gault or 24-hour creatinine clearance collection)
6. PT/INR <1.5 x ULN and PTT/ aPTT <1.5 x ULN

Exclusion Criteria:

1. Mixed small cell and NSCLC histology
2. A history of CNS involvement except as follows: Subjects with previously treated CNS metastases that are adequately treated with whole brain radiotherapy, that are neurologically stable, and do not require corticosteroids for symptomatic management for at least 14 days prior to first dose of study drug. There must be no clear evidence of radiographically active disease for at least 90 days prior to enrollment.
3. Anti-tumor therapy within 21 days of study Day 1
4. Prior treatment with ibrutinib or other BTK inhibitor anti-CD137 or CTLA-4 antibody. The following are exceptions to this criterion: Subjects previously treated with an anti-PD1, anti-PD-L1, or anti-PD-L2 antibody.
5. History of allogeneic organ transplant
6. Treatment with a strong cytochrome P450 (CYP) 3A inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaiah Dimery, Study Director — Pharmacyclics LLC.
Locations (16):
- United States (16):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - San Francisco, California
  - Gainesville, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - Hackensack, New Jersey
  - Durham, North Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b: In the Phase 1b (safety portion) of the study, a starting dose of 560 mg of ibrutinib and 10 mg/kg of MEDI4736 will be explored and will follow a 6 + 3 dose de-escalation design and will include a sentinel participant which will have a 3-day observation period prior to dosing of subsequent participants. Participants with one of the following three tumor types will be eligible for enrollment: NSCLC (adenocarcinoma and squamous-cell carcinoma), breast cancer (triple-negative and HER2-positive cancer), and Pancreatic cancer (adenocarcinoma).
Period: Period 1
Arm/Group | Phase 1b | Phase 2
Started | 7 (All Phase 1b participants went on to participate in Phase 2.) | 0
Completed | 6 | 0
Not Completed | 1 | 0
Not completed — Other varied reasons | 1 | 0
Period: Period 2
Arm/Group | Phase 1b | Phase 2
Started | 0 | 124 (Phase 2 includes all subjects who participated in Phase 1b.)
Completed | 0 | 0
Not Completed | 0 | 124
Not completed — Withdrawal by Subject | 0 | 14
Not completed — Death | 0 | 84
Not completed — Lost to Follow-up | 0 | 2
Not completed — Study Terminated by Sponsor | 0 | 14
Not completed — Other varied reasons | 0 | 10

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes all patients that received at least one dose of study treatment.
Groups:
- Phase 1b/2: All participants who received at least one dose of study treatment.
Arm/Group | Phase 1b/2
Number analyzed (Participants) | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 116
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 104
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Ibrutinib and Durvalumab (MEDI4736) and to Find the Recommended Phase II Dose.
Time Frame: From the date of first study treatment until DLT or disease progression per RECIST 1.1.
Measure: Number; unit: participants
Arm/Group | Phase 1b
Number analyzed (Participants) | 6
participants | 6

2. Primary Outcome: Phase 2: Efficacy of Ibrutinib in Combination With Durvalumab (MEDI4736) in Participants With Relapsed or Refractory Solid Tumors by Assessing the ORR Per RECIST 1.1.
Time Frame: From the date of first study treatment until progressive disease per RECIST 1.1 or unacceptable toxicity.
Population: The Response-evaluable population was participants who received at least 1 dose of treatment (ibrutinib and durvalumab) and provided 1 post-baseline response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 105
Participants | 2

3. Secondary Outcome: Phase 1b/2: Pharmacokinetics (Cmax) of Ibrutinib
Description: Cmax = the peak (maximum) plasma concentration of ibrutinib during the dosing interval on Cycle 3 Day 1.
Time Frame: 0hr, 1hr, 2hr, and 4hr post-dose
Population: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data. Data were analyzed together for Phase 1b and Phase 2 because the dose was the same.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase 1b/2 (Pharmacokinetic Population): All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Arm/Group | Phase 1b/2 (Pharmacokinetic Population)
Number analyzed (Participants) | 34
ng/mL | 218 (163)

4. Secondary Outcome: Phase 1b/2: Pharmacokinetics (AUC0-24h) of Ibrutinib
Description: AUC0-24 = the area under the plasma concentration-time curve of ibrutinib during the dosing interval on Cycle 3 Day 1
Time Frame: 0hr, 1hr, 2hr, and 4hr post-dose
Population: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data. Data were analyzed together for Phase 1b/2 because the dose was the same.
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Phase 1b/2 (Pharmacokinetic Population)
Number analyzed (Participants) | 34
h.ng/mL | 2126 (1315)

5. Secondary Outcome: Phase 1b/2: Pharmacokinetics (Cmax) of Durvalumab (MEDI4736)
Description: Cmax = the peak (maximum) plasma concentration of durvalumab (MEDI4736) after administration on Cycle 6 Day 1.
Time Frame: 60 minutes post-dose (dose administered as an infusion over a 1 hour period)
Population: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase 1b/2 (Pharmacokinetic Population)
Number analyzed (Participants) | 8
μg/mL | 386 (19.5)

6. Secondary Outcome: Phase 1b/2: Pharmacokinetics (Ctrough) of Durvalumab (MEDI4736)
Description: Ctrough = the trough plasma concentration of durvalumab (MEDI4736) after administration on Cycle 6 Day 1
Time Frame: Pre-dose
Population: All participants who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase 1b/2 (Pharmacokinetic Population)
Number analyzed (Participants) | 10
μg/mL | 168 (19.6)

7. Secondary Outcome: Phase 1b: Pharmacodynamics
Description: BTK occupancy
Time Frame: From the date of first study treatment until DLT or disease progression per RECIST 1.1.
Population: Data not collected
Arm/Group | Phase 1b
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 2: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Ibrutinib and Durvalumab (MEDI4736)
Time Frame: From the date of first study treatment until DLT or disease progression per RECIST 1.1.
Population: Participants who enrolled and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2
Number analyzed (Participants) | 122
Participants | 122

9. Secondary Outcome: Phase 2: Pharmacodynamics
Description: BTK binding site occupancy of ibrutinib was measured from peripheral blood samples collected from participants during Cycle 3 Day 1.
Time Frame: Pre-dose
Population: All subjects who received at least one dose of ibrutinib and who had at least one evaluable BTK occupancy assay result at Cycle 3 Day 1.
Measure: Mean (Standard Error); unit: percentage of BTK binding site occupancy
Arm/Group | Phase 2
Number analyzed (Participants) | 30
percentage of BTK binding site occupancy | 87.8 (4.2)

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Description: Adverse events were not collected by phase (Arm) because the treatments between Phase 1b and Phase 2 were not appreciably different.
Groups:
- Phase 1b/2: All subjects who received at least one dose of study treatment.
Arm/Group | Phase 1b/2
All-Cause Mortality (participants affected / at risk) | 96/122
Serious Adverse Events (participants affected / at risk) | 77/122
Other Adverse Events (participants affected / at risk) | 122/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b/2 (N=122)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Supraventricular tachycardia (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 6
Death (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 2
Asthenia (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Pneumonia (Hepatobiliary disorders) | 8
Sepsis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Serratia bacteraemia (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Embolic stroke (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 8
Stenotrophomonas sepsis (Infections and infestations) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b/2 (N=122)
Anaemia (Blood and lymphatic system disorders) | 26
Nausea (Gastrointestinal disorders) | 33
Diarrhoea (Gastrointestinal disorders) | 22
Abdominal pain (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 19
Stomatitis (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 53
Oedema peripheral (General disorders) | 26
Pyrexia (General disorders) | 19
Urinary tract infection (Infections and infestations) | 8
Aspartate aminotransferase increase (Investigations) | 15
Weight decreased (Investigations) | 12
Alanine aminotransferase increased (Investigations) | 11
Blood alkaline phosphatase increased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 28
Hyponatraemia (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 19
Pruritus (Skin and subcutaneous tissue disorders) | 14
Rash erythematous (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT02403271/SAP_000.pdf
  • Study Protocol (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT02403271/Prot_001.pdf